CLINICAL TRIAL: NCT00384436
Title: Fixed Dose Comparison of Escitalopram to an Active Comparator in Severely Depressed Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT-MD-39
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of escitalopram to an active comparator in severely depressed patients

DETAILED DESCRIPTION:
Escitalopram is the S-enantiomer of citalopram. Both escitalopram and citalopram are selective serotonin reuptake inhibitors (SSRIs) and are used to treat depression in adults. This study is designed to evaluate the safety and efficacy of escitalopram and an active comparator in severely depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet DSM-IV criteria for Major Depressive Disorder.
* Patients must have severe depression.
* MADRS greater than or equal to 30

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control.
* Patients who are considered a suicide risk.
* Patients who currently meet DSM-IV criteria for: a principal diagnosis for Axis I disorder other than MDD (comorbid GAD is allowed), bipolar disorder, schizophrenia or any psychotic disorder, obsessive-compulsive disorder, dysthymia.
* Patients with a family history of bipolar disorder, schizophrenia, or any psychotic disorder.
* Patients with history of any psychotic disorder or any psychotic feature.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time to premature discontinuation

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS)

CONTACTS AND LOCATIONS:
Locations (1):
- For information regarding investigative sites, contact Forest Professional Affairs, St Louis, Missouri, United States

REFERENCES:
- [Derived] Bose A, Tsai J, Li D. Early non-response in patients with severe depression: escitalopram up-titration versus switch to duloxetine. Clin Drug Investig. 2012 Jun 1;32(6):373-85. doi: 10.2165/11631890-000000000-00000. PMID 22559255
- [Derived] Signorovitch J, Ramakrishnan K, Ben-Hamadi R, Yu AP, Wu EQ, Dworak H, Erder MH. Remission of major depressive disorder without adverse events: a comparison of escitalopram versus serotonin norepinephrine reuptake inhibitors. Curr Med Res Opin. 2011 Jun;27(6):1089-96. doi: 10.1185/03007995.2011.567255. Epub 2011 Mar 28. PMID 21438794